CLINICAL TRIAL: NCT02400359
Title: Lorcaserin in Obesity: Identification of CNS Targets Using FMRI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P000196
Record Dates: First submitted 2015-01-12; First posted 2015-03-27 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Weight Loss
Keywords: fMRI; Magnetic Resonance Imaging; endocrinology; MRI; obesity; weight loss; lorcaserin
MeSH Terms: conditions — Obesity; Weight Loss | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be randomized to either placebo or Lorcaserin HCl.
  Interventions: Drug: Placebo
- Active (Active Comparator): Subjects will be randomized to either placebo or Lorcaserin HCl.
  Interventions: Drug: Lorcaserin HCl

INTERVENTIONS:
Drug: Lorcaserin HCl — Lorcaserin is a weight-loss drug developed by Arena Pharmaceuticals. It has serotonergic properties and acts as an anorectic.
  Other Names: Belviq
  Arms: Active
Drug: Placebo — This is a placebo oral pill that is a visual replica of the Lorcaserin medication but with no active ingredients.
  Arms: Placebo

SUMMARY:
The purpose of this protocol is to investigate, using functional magnetic resonance imaging (fMRI), the effect of treatment with lorcaserin on centers of the brain that control appetite and food intake, as well as lorcaserin's downstream metabolic effects.

DETAILED DESCRIPTION:
The purpose of this protocol is to investigate the effect of treatment with the study drug, called lorcaserin on centers of the brain that control appetite and food intake, as well as lorcaserin's other metabolic effects. Lorcaserin's effect on the brain will be investigated using functional magnetic resonance imaging (fMRI). Lorcaserin was approved in June 2012 as an addition to a reduced-calorie diet and exercise, for chronic weight management. Previous weight loss drugs, such as fenfluramine, acted throughout the body and caused heart problems. Lorcaserin is different because it only acts on receptors (sites of action) that are found in the brain and does not act on the heart, and thus, has not been shown to cause the heart problems seen in the past.

1. To examine the effects of the study drug lorcaserin, on the brain, and its impact on food visualization (high fat and low fat images) and interaction with satiety (by measuring during the fasting or fed states) using fMRI. (Satiety is defined as when a person has had enough or too much food and does not want to eat any more, as after finishing a satisfying meal.)
2. To examine the satiety and weight-reducing effect of lorcaserin using physiological measurements (such as how much weight is lost and how this may affect hormone levels), and its association with changes in fMRI responses and neuropsychological performance. To examine whether the long-term weight reducing effects of lorcaserin can be predicted by early food visualization.

ELIGIBILITY:
Inclusion Criteria:

Obese: BMI> 30 kg/m2 or >27 kg/m2 with comorbidities (including but not limited to insulin resistance, hypertension, dyslipidemia, cardiovascular disease, stroke, sleep apnea, gallbladder disease, hyperuricemia and gout, and osteoarthritis).

Additionally, women participants must use double barrier methods to prevent pregnancy (diaphragm with intravaginal spermicide, cervical cap, male or female condom with spermicide). If a woman suspects that she has become pregnant at any time or does not use one of the contraceptive methods recommended by the investigator, she must notify the study staff. If a woman becomes pregnant, she will be withdrawn from the study. The study staff will follow the progress of her pregnancy and the birth of her child.

Exclusion Criteria:

1. Subjects using any other weight loss products (orlistat, phentermine, topiramate, fenfluramine, dexfenfluramine, amphetamines, GLP-1 agonists) or use within 3 months.
2. Women who are breastfeeding, pregnant, or wanting to become pregnant.
3. Women using IUD (intrauterine device)
4. Any change in the dosage of hormonal contraceptive medications (birth control pills, implanon). Subjects should remain on same medication/ same dose during the time of the entire study.
5. Moderate (creatinine clearance of 30-59 ml/min) and severe renal impairment (creatinine clearance below 30 ml/min) and end-stage renal disease
6. Moderate, or severe hepatic impairment
7. Hypersensitivity to the active substance or any of the excipients in lorcaserin
8. Congestive heart failure and/or pulmonary hypertension
9. Arrhythmias (bradycardia, tachycardia) and valvular heart diseases
10. Diagnosis of diabetes, defined per ADA criteria as Hba1c > 6.5% and/or fasting glucose > 125 mg/dL and/or random glucose > 200 mg/dL
11. Inflammatory conditions like inflammatory bowel disease, Rheumatoid arthritis etc.
12. Alcohol consumption- the maximum quantity for men is 140g-210g per week. For women, the range is 84g-140g per week or drinking as consuming no more than two drinks a day for men and one for women. Alcohol can cause increased risk of pancreatitis and hypoglycemia.
13. Untreated thyroid disease like hypothyroidism or hyperthyroidism
14. Subjects taking the following medications: phosphodiesterase inhibitors, serotonergic medications (e.g. SSRI (selective serotonin reuptake inhibitor), SNRI, MAO (monoamine oxidase) inhibitors, bupropion, tricyclic antidepressants, St. John's Wort), valproic acid, codeine (CYP2D6 inhibition), tamoxifen, timolol, warfarin, steroids (inhaled or systemic due to reduced hypoglycemic effect), and subjects on other hormones (LHRH analogs etc).
15. Subjects with any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g. cochlear implants, pacemakers, neuron or biostimulators, electronic infusion pumps, etc.)
16. Subjects with any type of metallic implant that could potentially be displaced or damaged during MRI, such as aneurysm clips, metallic skull plates, surgical implants etc. or metal containing tattoos
17. Anxiety of small spaces and/or claustrophobia
18. Uncontrolled cardiac impairment, circulatory impairment, or inability to perspire (poor thermoregulatory function)
19. Significant sensory or motor impairment
20. Epilepsy, particularly photo-sensitive epilepsy, which may place the individual at a higher risk for adverse events during fMRI scanning with visual stimulation
21. Subjects with neurological problems which may interfere with or complicate testing (e.g. presence of titubation)
22. Body weight above the limitation of the MRI scanning table (330lbs/150 Kg) or body dimensions that could difficult the performance of the scan.
23. Subjects who cannot adhere to the experimental protocol for any reason
24. Anemia with Hgb less than 10
25. Uncontrolled infectious diseases (e.g. HIV, hepatitis, chronic infections etc)
26. Any uncontrolled endocrine condition, e.g. Cushing's, Acromegaly, etc
27. Any cancers or lymphoma
28. Eating disorders like anorexia, bulimia
29. Weight loss surgery or gastrectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
fMRI (Functional changes in the brain) | 28 days

SECONDARY OUTCOMES:
Body Composition (DEXA) | 6 months
  Changes in body composition will be assessed by the following measurements:
  DEXA (Dual Energy X-Ray Absorptiometry): Body composition and bone density will be measured by DEXA. For the DEXA test, the subject will be lying on an examination bed for about 25 minutes. A small part of the DEXA machine will be recording and moving back and forth about 3 feet above their body. The radiation the subject will get is very small and is much less than what one gets from a regular chest X-Ray.
  Anthropometry: Anthropometry will be performed by a licensed dietician. Measurements include: Height, Weight, umbilical and smallest waist, broadest and iliac hip measurements.
Metabolic Rate (Resting Metabolic Rate (RMR) | 6 months
  Resting Metabolic Rate (RMR): RMR is the amount of calories the subject burn without doing any physical work. The subject's RMR will be measured with a commonly used instrument. The subject will be asked to lie quietly in bed and stay awake with a large plastic hood over the subject's head and upper body for about 20 minutes. The subject will breathe normally while the air they breathe out is collected and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Christos S Mantzoros, MD DSc, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farr OM, Upadhyay J, Gavrieli A, Camp M, Spyrou N, Kaye H, Mathew H, Vamvini M, Koniaris A, Kilim H, Srnka A, Migdal A, Mantzoros CS. Lorcaserin Administration Decreases Activation of Brain Centers in Response to Food Cues and These Emotion- and Salience-Related Changes Correlate With Weight Loss Effects: A 4-Week-Long Randomized, Placebo-Controlled, Double-Blind Clinical Trial. Diabetes. 2016 Oct;65(10):2943-53. doi: 10.2337/db16-0635. Epub 2016 Jul 6. PMID 27385157